CLINICAL TRIAL: NCT03566966
Title: Clinical Relevance of Serum Non-organ-specific Antibodies in Hepatitis C Virus Patients Receiving Direct-acting Antiviral Therapy
Brief Title: Autoantibodies and Direct-acting Antivirals
Acronym: BIOEPA
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Clinical professor, University of Bari
Other Study IDs: Policlinic Hospital 3, Bari
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Viral Hepatitis C; Therapy Adverse Effect
Keywords: hepatitis C virus infection; non-organ-specific antibodies; prognostic value; sustained virological response
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Biospecimen Retention: Samples Without DNA — Serum samples for antibodies determination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-organ-specific Ab positive: Patients who had detectable circulating autoantibodies before treatment with antivirals.
  Interventions: Biological: Non-organ-specific Ab positive
- Non-organ-specific Ab negative: Patients who did not have detectable circulating autoantibodies before treatment with antivirals.
  Interventions: Biological: Non-organ-specific Ab negative

INTERVENTIONS:
Biological: Non-organ-specific Ab positive — Antiviral administration and evaluation of SVR24 and side effects
  Other Names: direct-acting antiviral agents
  Groups: Non-organ-specific Ab positive
Biological: Non-organ-specific Ab negative — direct-acting antiviral agents
  Groups: Non-organ-specific Ab negative

SUMMARY:
The investigators assessed non-organ-specific antibodies before and 24 weeks after the end of therapy with direct-acting antivirals, in order to better clarify the clinical relevance of these antibodies in terms of treatment response and prognostic value.

To achieve this goal patients with hepatitis C virus related advanced liver disease, with detectable circulating autoantibodies on at least two determinations before treatment, were enrolled.

DETAILED DESCRIPTION:
About 40-70% of hepatitis C virus patients develop at least an autoimmune extra-hepatic disorder presumably due to the interaction between hepatitis C virus E2 envelope protein and B lymphocyte Cluster of Differentiation-81 receptor. In addition, the same interaction is responsible for the production of different serum non-organ-specific antibodies. The clinical significance of the latter phenomenon has not been fully understood except for the presence of liver kidney microsome-1 antibody, which is linked to a molecular mimicry between the cytochrome enzyme CYP2D6, primarily expressed in the liver, and hepatitis C virus proteins in genetically predisposed subjects.

Actually, no data are available about the prevalence and clinical significance of serum non-organ-specific antibodies in hepatitis C virus patients treated with second generation direct-acting antivirals.

ELIGIBILITY:
Inclusion Criteria:

HCV positive patients Presence of advanced liver fibrosis Eligibility to the treatment with direct-acting antiviral therapy.

Exclusion Criteria:

History of autoimmune hepatitis and/or cholangitis Evidence of active hepatocellular carcinoma Human immunodeficiency virus coinfection Hepatitis B virus coinfection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caucasian patients affected by chronic hepatitis C virus infection who were consecutively admitted as outpatients to the Gastroenterology Unit, Policlinic Hospital, Bari, Italy, from July 2015-August 2016 to receive a treatment with second generation direct-acting antivirals.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks after the end of antiviral therapy
  Evaluation of HCV-RNA levels

SECONDARY OUTCOMES:
Disappearance of non-organ-specific antibodies | 24 weeks after the end of antiviral therapy
  Evaluation of anti nuclear antibodies, anti smooth muscle antibodies, liver kidney microsome antibodies
Side effects | 24 weeks after the end of antiviral therapy
  Clinical manifestations and laboratory alterations

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Di Leo, MD, PhD, Study Chair — University of Bari
Locations (1):
- Policlinic Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It depends on the possibility to merge similar data and produce a multicentric study

REFERENCES:
- [Derived] Shahini E, Iannone A, Romagno D, Armandi A, Carparelli S, Principi M, Viggiani MT, Ierardi E, Di Leo A, Barone M. Clinical relevance of serum non-organ-specific antibodies in patients with HCV infection receiving direct-acting antiviral therapy. Aliment Pharmacol Ther. 2018 Nov;48(10):1138-1145. doi: 10.1111/apt.14999. PMID 30375693